CLINICAL TRIAL: NCT00112086
Title: Feasibility Study of Neoadjuvant Chemotherapy Followed by Interval Cytoreductive Surgery for Stage III/IV Ovarian, Tubal and Peritoneal Cancers: JCOG0206
Brief Title: OVCA-NAC-P2: Study of Chemotherapy Followed by Cytoreductive Surgery for Ovarian, Tubal and Peritoneal Cancers: JCOG0206
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Hiroyuki Yoshikawa , MD, Study Chair, Japan Clinical Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0206; C000000005
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: ovarian neoplasms; laparoscopy; neoadjuvant therapy; interval cytoreductive surgery
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — Neoadjuvant Therapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy (Paclitaxel and Carboplatin)

SUMMARY:
A feasibility study of neoadjuvant chemotherapy (NAC) followed by interval cytoreductive surgery (ICS) and postoperative chemotherapy for stage III/IV mullerian carcinomas such as ovarian, tubal and peritoneal carcinomas.

DETAILED DESCRIPTION:
The purposes are to assess the safety and efficacy of the treatment starting with NAC and to know whether we can accurately diagnose these advanced carcinomas by imaging studies, cytologic findings and tumor markers without staging laparotomy or laparoscopy. Fifty-six patients with advanced mullerian carcinomas will be recruited to the study. After confirmation of diagnosis by laparoscopic inspection and biopsies, patients undergo 4 cycles of chemotherapy as NAC followed by ICS and additional 4 cycles of postsurgical chemotherapy. The primary endpoint is proportion of clinical complete remission after accomplishment of the protocol treatment and the major secondary endpoint is positive predictive value of diagnosis before laparoscopy regarding tumor origin, histology and stage. Based on the result of this study, we will conduct a phase III study to compare the treatment starting with NAC and primary cytoreductive surgery followed by postsurgical chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV müllerian carcinoma by prelaparoscopic clinical findings including imaging studies (CT, MRI or ultrasonography)
* Cytology of ascites, pleural effusions, or fluids obtained by tumor centesis
* Malignancies of other origins, such as breasts and digestive tract, should be excluded by endoscopy, opaque enema, or ultrasonography when these malignancies are suspected from symptoms, physical examinations or imaging diagnosis.
* CA125>200U/ml and CEA<20ng/ml.
* Clinically deemed to be a candidate for debulking surgery without evidence of brain, bone, bone marrow metastases, multiple lung, or multiple liver metastases
* Presence of at least one measurable lesion
* Previously untreated for these malignancies and no history of treatment with chemotherapy or radiotherapy even for other diseases
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3,
* Adequate bone marrow, hepatic, renal, cardiac and respiratory functions, and
* Written informed consent.

Exclusion Criteria:

* Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ
* Pregnant or nursing
* Severe mental disorders
* Systemic and continuous use of steroidal drugs
* Active infections
* Uncontrolled hypertension
* Diabetes mellitus, uncontrolled or controlled with insulin
* History of cardiac failure, unstable angina, myocardial infarction within 6 months prior to the registration
* Liver cirrhosis or bleeding tendency contraindicating debulking surgery
* Intestinal occlusion necessary for surgical treatment
* Hypersensitivity to alcohol

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
proportion of clinical complete remission

SECONDARY OUTCOMES:
positive predictive value (PPV) of prelaparoscopic diagnosis concerning the origin and histology
proportion of the patients diagnosed as müllerian carcinoma by laparoscopic inspection and histopathology of biopsy specimen among those diagnosed by prelaparoscopic findings
PPV of prelaparoscopic diagnosis concerning clinical stage; proportion of the patients diagnosed as stage III or IV by laparoscopic inspection among those diagnosed by prelaparoscopic findings
PPV of overall prelaparoscopic diagnosis; proportion of the patients diagnosed as stage III or IV müllerian carcinoma by laparoscopic inspection and histopathology of biopsy specimen among those diagnosed by prelaparoscopic findings
response rate to NAC among patients whose clinical diagnosis is confirmed by laparoscopy
proportion of patients who received interval cytoreductive surgery (ICS) among patients whose clinical diagnosis is confirmed by laparoscopy
progression-free survival among patients whose clinical diagnosis is confirmed by laparoscopy
operative morbidity among all enrolled patients
adverse events among all enrolled patients, and
overall survival among all enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Yoshikawa, MD, Study Chair — University of Tsukuba
Locations (1):
- National Cancer Center, Tsukiji, 5-1-1, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Background] Onda T, Kamura T, Ishizuka N, Katsumata N, Fukuda H, Yoshikawa H; Japan Clinical Oncology Group Study JCOG0206. Feasibility study of neoadjuvant chemotherapy followed by interval cytoreductive surgery for stage III/IV ovarian, tubal and peritoneal cancers: Japan Clinical Oncology Group Study JCOG0206. Jpn J Clin Oncol. 2004 Jan;34(1):43-5. doi: 10.1093/jjco/hyh007. PMID 15020662
- [Derived] Onda T, Kobayashi H, Nakanishi T, Hatae M, Iwasaka T, Konishi I, Shibata T, Fukuda H, Kamura T, Yoshikawa H. Feasibility study of neoadjuvant chemotherapy followed by interval debulking surgery for stage III/IV ovarian, tubal, and peritoneal cancers: Japan Clinical Oncology Group Study JCOG0206. Gynecol Oncol. 2009 Apr;113(1):57-62. doi: 10.1016/j.ygyno.2008.12.027. Epub 2009 Jan 31. PMID 19181369
- See also: Related Info — http://www.jcog.jp/